CLINICAL TRIAL: NCT01349205
Title: Caffeine in Children With Obstructive Sleep Apnea, Dose Response Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study medication was no longer available in the market
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Memorial Hermann Hospital (Other)
Responsible Party: Principal Investigator, Samia Khalil, Professor - Anesthesiology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-09-0457; HSC-MS-09-0457 (Other: Memorial Hermann CPHS)
Record Dates: First submitted 2011-05-03; First posted 2011-05-06 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Obstructive Sleep Apnea; Enlargement of Tonsil or Adenoid
Keywords: OSA; Caffeine; Tonsillectomy; Adenoidectomy; Sleep Study
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Caffeine; Sodium Benzoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Caffeine and Sodium Benzoate 10 mg/kg IV (Experimental): Group 1 of randomized study.
  Interventions: Drug: Caffeine and sodium Benzoate 10 mg/kg IV
- Caffeine and Sodium Benzoate 20 mg/kg IV (Experimental): Group 2 of randomized study
  Interventions: Drug: Caffeine and Sodium Benzoate 20 mg/kg IV
- 0.9 NS Saline (Placebo Comparator): Control group of randomized study.
  Interventions: Drug: 0.9 NS Saline

INTERVENTIONS:
Drug: Caffeine and sodium Benzoate 10 mg/kg IV — IV, 10mg/kg, IVP, 1 time
  Arms: Caffeine and Sodium Benzoate 10 mg/kg IV
Drug: Caffeine and Sodium Benzoate 20 mg/kg IV — IV, 20 mg/kg, IVP, 1 time
  Arms: Caffeine and Sodium Benzoate 20 mg/kg IV
Drug: 0.9 NS Saline — IV, 0-10 ml, IVP, 1 time
  Arms: 0.9 NS Saline

SUMMARY:
The aim of this study is to evaluate whether a smaller dose of caffeine sodium benzoate 10 mg/kg IV is as effective as 20 mg/kg IV in decreasing the number of children who develop post extubation adverse upper airway respiratory events compared to placebo.

DETAILED DESCRIPTION:
Institutional approval and written informed consent from parents or guardians of healthy children, with obstructive sleep apnea (OSA) and/or with increased end-tidal C02 (sleep related hypoventilation, obstructive hypoventilation or sustained alveolar hypoventilation), confirmed with sleep study, scheduled for elective outpatient or inpatient adeno-tonsillectomy at our hospital, will be obtained. The study will be prospective, randomized, double blinded and placebo controlled. A computer generated randomization list will be used, and the study will be registered with clinical.trials.gov. Written child assent will be obtained from children 7 years and older. Copies of a flyer and an explanation of the study will be provided at the office of all the pediatric ENT surgeons who practice at the Memorial Hermann Hospital OR. The investigators will communicate with the nurses at the surgeons' office and ask them to give the flyer with an explanation of the study to the parents and children on the day they schedule the surgery. The flyer with an explanation of study will be sent to IRB for review and approval. A research assistant will invite parents or guardians in the DSU unit, anesthesia clinic or on the floor to allow their children to be part of the study. Children with OSA and/or increased end tidal C02 (sleep related hypoventilation, obstructive hypoventilation or sustained alveolar hypoventilation), 2-12 years of age, and both genders will be eligible to be part of the study. OSA and its severity will be diagnosed by a preoperative polysomnography. Children with compromised cardiovascular, pulmonary or renal function, those with congenital syndromes, sickle cell disease, history of seizures and those receiving theophylline will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Children with OSA and/or increased end tidal C02 (sleep related hypoventilation, obstructive hypoventilation or sustained alveolar hypoventilation), 2-12 years of age, and both genders will be eligible to be part of the study. OSA and its severity will be diagnosed by a preoperative polysomnography.

Exclusion Criteria:

* Children with compromised cardiovascular, pulmonary or renal function, those with congenital syndromes, sickle cell disease, history of seizures and those receiving theophylline will be excluded.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2010-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Effects of Caffeine | Immediately after drug administration upto 24 hours
  The primary outcome of the study is the number of children who develop adverse postextubation respiratory events, including: 1) airway obstruction, requiring jaw-chin thrust maneuver, or placement of an LMA or endotracheal tube, 2) laryngospasm, requiring continuous positive airway pressure or intervention with a muscle relaxant, 3) apnea, 4) desaturation(defined as a decrease in oxygen saturation <95% while breathing oxygen via mask which is our hospital and PACU nurses standard of care), 5) hypoventilation/ hypercapnia )

SECONDARY OUTCOMES:
Caffeine Drug Effects | Immediately after drug administration to 24 hours
  A secondary outcome of the study will be the incidence of adverse post-extubation respiratory events.

CONTACTS AND LOCATIONS:
Overall Officials: samia Khalil, MD, Principal Investigator — Memorial Hermann Hospital
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States